CLINICAL TRIAL: NCT06505096
Title: A Comparative Study of the Results of Dynamic and OPD Static Measurement of Pupil Diameter Before and After Cataract Surgery by Pupil Detectors
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Other Study IDs: QX-2023-A-012
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Cataract
Keywords: cataract; pupil size
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Orthokeratology group: -0.5D~+0.0D
  Interventions: Procedure: cataract surgery
- myopia group: SE lens less than -0.5D
  Interventions: Procedure: cataract surgery
- hyperopia group: SE more than +0.5D
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — Phaco+IOL implention

SUMMARY:
Age-related cataract remains the leading cause of blindness in developing countries. And, with the aging of the population in these countries, the number of cataract patients will continue to grow. With accurate biological measurements and the implantation of a suitable IOL, most cataract patients can achieve good distance vision after surgery. Studies have shown differences in pupil diameter and sensitivity in patients with different refractive states, with correlations to accommodation status as well as refractive error. The pupil is an important factor to be evaluated during the selection of an artificial lens (Intraocular lens, IOL), especially a functional IOL.

Among the various instruments used for preoperative cataract biological measurements, the light source is mostly a fixed parameter, and the static pupil diameter measurement by fixed illumination light source detection as an evaluation method is relatively rough. In this study, we are going to simulate different illumination states in daily life and set up two kinds of measurement instruments, namely, OPD and binocular pupil detector, so as to obtain more realistic research results and to explore the following: 1. The static and dynamic measurement of pupil diameter by people of different refractive states in different periods of preoperative and postoperative period. 2. Whether there is a difference between the static and dynamic pupil measurement results, 2. the change of pupil size under the stimulation of different light sources, and to compare the difference between the two detection methods, to provide objective pupil indexes for the more scientific selection of functional IOLs, to provide a basis for the selection of more accurate pupil measurement methods, to accurately screen the population of the use of functional IOLs, and to improve the patient's satisfaction after the operation.

Purpose of the study To simulate the difference between the preoperative and postoperative pupil diameters of cataract patients measured by static and dynamic methods under daily illumination, to select a more accurate pupil measurement method, and to make corrections for the evaluation of preoperative biometric indexes.

ELIGIBILITY:
Inclusion Criteria:

(1) diagnosed with cataract; (2) treated with lens ultrasonic emulsification combined with monofocal IOL implantation in our hospital; (3) agreed to participate and cooperate with this study.

Exclusion Criteria:

(1) acute eye disease symptoms, such as eye redness, eye pain, increased ocular secretions, etc.; (2) other eye diseases that seriously affect visual function in both eyes, such as amblyopia, high myopia, glaucoma, diabetic retinopathy, severe age-related macular degeneration and retinal detachment, etc.; (3) intra-operative or post-operative complications in cataract surgery; combined with other ophthalmic surgeries; and any other ophthalmic surgery for both eyes in the follow-up period; the presence of any other ophthalmic surgery in both eyes in the follow-up period. (4) Inability to understand the informed consent form and inability to communicate.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty eyes of patients who were treated with lens ultrasonic emulsification combined with IOL implantation in our hospital were selected. According to the preoperative refractive status, they were divided into orthokeratology group (-0.5D~+0.5D), myopia group less than -0.5D, hyperopia group more than +0.5D, 20 eyes in each group.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
pupil size | 1 week, 1 month, 3 months
  pupil size before and after cataract surgery

IPD SHARING:
Plan to Share IPD: No